CLINICAL TRIAL: NCT05065931
Title: Real-world Effectiveness Evaluation of Clinical Decision Support System Based on Artificial Intelligence (AI-CDSS) on Diagnosis
Brief Title: Real-world Effectiveness Evaluation of Clinical Decision Support System Based on Artificial Intelligence (AI-CDSS)
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 324-01
Record Dates: First submitted 2019-07-12; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2019-07

CONDITIONS: Medical Informatics Applications

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before: before CDSS on-line
- After: after CDSS on-line
  Interventions: Other: Auxiliary diagnostic system by AI-CDSS

INTERVENTIONS:
Other: Auxiliary diagnostic system by AI-CDSS — Helping clinicians to make diagnoses by using CDSS based-on AI
  Groups: After

SUMMARY:
This study intends to explore the accuracy of clinical diagnosis of AI based CDSS system and promotion of clinical work by comparing CDSS before and after the online.

DETAILED DESCRIPTION:
This study intends to explore the accuracy of clinical diagnosis of AI based CDSS system and promotion of clinical work by comparing CDSS before and after the online. The difference of diagnostic accuracy before and after AI-CDSS application will be compared by the before and after design, and the role of AI-CDSS will be explored.

ELIGIBILITY:
Inclusion Criteria:

* all hospitalized patients in 6 clinical departments, Otolaryngology, Orthopaedic, Respiratory Medicine, General Surgery, Cardiology and Hematology from December 2016 to February 2019.

Exclusion Criteria:

* Missing data for key variables

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population was the hospitalized patient from December 2016 to February 2019 in 6 clinical departments. The six clinical departments were Otolaryngology, Orthopaedic, Respiratory Medicine, General Surgery, Cardiology and Hematology.
Sampling Method: Non-Probability Sample
Enrollment: 34113 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Accuracy Rate of Recommended Diagnosis by CDSS, up to 12 weeks | When the subject was discharged from the hospital
  Based on the patient's discharge diagnosis as a standard, it is explored whether the diagnosis given by the CDSS is consistent with the discharge diagnosis in the patient's medical record.
Patients' hospitalization time (days), up to 24 weeks | When the subject was discharged from the hospital
  The length of a patient's stay is the number of days he or she experiences from the time of admission to the time of discharge.
consistency between admission diagnosis and discharge diagnosis up to 12 weeks | When the subject was discharged from the hospital
  When the patient comes to the hospital, the clinician will write an inpatient record and give a preliminary diagnosis, which we call admission diagnosis.After the patient is hospitalized, all kinds of examinations will be improved. After all the examination results come out, the patient's diagnosis on admission may be modified. Because there are no auxiliary examination results on admission, the diagnosis on admission may not be completely correct.This modified diagnosis is called discharge diagnosis.This study compared the consistent rate of admission diagnosis and discharge diagnosis before and after CDSS on-line.

SECONDARY OUTCOMES:
length of confirmed time, up to 6 weeks | When the subject was discharged from the hospital
  he length of confirmed time (days) was the duration between the preliminary admission diagnosis and the definite diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, Ph.D, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
After the results of the study are published for one year, the data can be published to other researchers. But the data needs to be de-identified to protect the patient's privacy.